CLINICAL TRIAL: NCT00422968
Title: PREmier of Randomized COMparison of Bypass Surgery Versus AngioplasTy Using Sirolimus-Eluting Stent in Patients With Left Main Coronary Artery Disease
Brief Title: Bypass Surgery Versus Angioplasty Using Sirolimus-Eluting Stent in Patients With Left Main Coronary Artery Disease
Acronym: PRECOMBAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, M.D., Ph.D., FACC, CardioVascular Research Foundation, Korea
Organization: CardioVascular Research Foundation, Korea (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0012
Record Dates: First submitted 2007-01-16; First posted 2007-01-17 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; Stent; Bypass surgery, coronary artery
MeSH Terms: conditions — Coronary Artery Disease | interventions — Percutaneous Coronary Intervention; Coronary Artery Bypass

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- coronary artery bypass graft (Active Comparator): coronary artery bypass graft
  Interventions: Procedure: coronary artery bypass graft
- percutaneous coronary intervention (Experimental): Using silorimus eluting stent
  Interventions: Device: Percutaneous coronary intervention

INTERVENTIONS:
Device: Percutaneous coronary intervention — Using silorimus eluting stent
  Arms: percutaneous coronary intervention
Procedure: coronary artery bypass graft — coronary artery bypass graft
  Arms: coronary artery bypass graft

SUMMARY:
The primary objective of the PRE-COMBAT trial is:

To establish the safety and effectiveness of coronary stenting with the sirolimus-eluting balloon expandable stent (Cordis Johnson & Johnson, Warren, New Jersey) compared with bypass surgery for the treatment of an unprotected LMCA stenosis. The alternative hypothesis is that the experimental strategy (coronary stenting with the sirolimus-eluting stents) is not inferior to the standard strategy (bypass surgery).

DETAILED DESCRIPTION:
Despite bypass surgery has been considered as the standard strategy for the treatment of unprotected left main coronary artery (LMCA) lesions, several studies have demonstrated that percutaneous coronary intervention (PCI) of the unprotected LMCA is feasible and appears to be an alternative strategy in selected patients. However, the safety and efficacy of PCI in patients with unprotected LMCA stenosis are still a matter of debate.

Previous studies have demonstrated the safety and feasibility of unprotected LMCA intervention using bare metal stents (BMS). There was a favorable initial outcome after LMCA intervention using BMS in low-risk patients. However, in-stent restenosis after BMS implantation has emerged as the interference to widely perform PCI for unprotected LMCA lesions and the most important reason for selection of bypass surgery as the first choice for treating LMCA stenosis. In-stent restenosis in these patients not only influences long-term survival, but also make repeat intervention more complex. Despite endeavors to decrease in-stent restenosis after LMCA intervention using BMS, such as aggressive debulking atherectomy, the restenosis rate still remains at 20-30%. The sirolimus-eluting stent (SES) (Cypher, Cordis, Johnson & Johnson Corp, Miami, Florida) markedly decreases in-stent restenosis in elective patients with relatively simple coronary lesions. In real-world practice using SES, patients undergoing SES implantation were treated with a less restrictive interventional approach. However, the results are very promising similar to the randomized controlled trials. These findings warrant new studies to compare the efficacy of SES for more complex lesion subsets including LMCA disease with coronary artery bypass graft (CABG).

ELIGIBILITY:
Inclusion Criteria:

* The patient must be at least 18 years of age.
* Significant de novo left main stenosis (>50% by visual estimation) with or without any additional target lesions (>70% by visual estimation)
* Left main lesion and lesions outside LMCA (if present) potentially equally treatable with coronary stenting and bypass surgery
* Patients with stable (CCS class 1 to 4) or acute coronary syndromes (unstable angina pectoris Braunwald class IB, IC, IIB, IIC, IIIB, IIIC or NSTEMI) or patients with atypical chest pain or without symptoms but having documented myocardial ischemia
* The patient or guardian agrees to the study protocol and the schedule of clinical and angiographic follow-up, and provides informed, written consent, as approved by the appropriate Institutional Review Board/Ethical Committee of the respective clinical site.

Exclusion Criteria:

* The patient has a known hypersensitivity or contraindication to any of the following medications:

  * Heparin
  * Aspirin
  * Both Clopidogrel and TIclopidine
  * Sirolimus, paclitaxel, ABT 578
  * Stainless steel and/or
  * Contrast media (patients with documented sensitivity to contrast which can be effectively pre-medicated with steroids and diphenhydramine [e.g. rash] may be enrolled. Patients with true anaphylaxis to prior contrast media, however, should not be enrolled).
* Systemic (intravenous) Sirolimus, paclitaxel or ABT-578 use within 12 months.
* Any previous PCI within 1 year
* Previous bypass surgery
* Any previous PCI of a LMCA or ostial left circumflex artery or ostial left anterior descending artery lesion within 1 year
* Intention to treat more than one totally occluded major epicardial vessel
* Acute MI patients within 1 week
* Patients with EF<30%.
* Patients with cardiogenic shock
* Any disabled stroke with neurological deficit or any cerebrovascular accident within 6 months
* Creatinine level > 2.0mg/dL or dependence on dialysis.
* Severe hepatic dysfunction (AST and ALT > 3 times upper normal reference values).
* Gastrointestinal or genitourinary bleeding within the prior 3 months, or major surgery within 2 months.
* History of bleeding diathesis or known coagulopathy (including heparin-induced thrombocytopenia), or will refuse blood transfusions.
* Current known current platelet count <100,000 cells/mm3 or Hgb <10 g/dL.
* An elective surgical procedure is planned that would necessitate interruption of thienopyridines during the first 1 year post enrollment.
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
* Patients who are actively participating in another drug or device investigational study, which have not completed the primary endpoint follow-up period.
* Subject unable or unwilling to follow-up with visits required by protocol
* Female of childbearing potential, unless a recent pregnancy test is negative, who possibly plan to become pregnant any time after enrollment into this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1454 (Actual)
Dates: Start 2005-03; Primary Completion 2009-11 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Major cardiac and cerebrovascular event (MACCE): the composite of death, myocardial infarction, stroke, and ischemica-driven target vessel revascularization | one-year after treatment

SECONDARY OUTCOMES:
All-cause mortality | at 30 days, 6 months, 1 year, and yearly to 5 years
Cardiac death | at 30 days, 6 months, 1 year, and yearly to 5 years
Myocardial infarction | at 30 days, 6 months, 1 year, and yearly to 5 years
Cerebrovascular accident | at 30 days, 6 months, 1 year, and yearly to 5 years
Target vessel revascularization (all and ischemia-driven) | at 30 days, 6 months, 1 year, and yearly to 5 years
Target lesion revascularization (all and ischemia-driven) | at 30 days, 6 months, 1 year, and yearly to 5 years
Stent thrombosis in the PCI group | at 30 days, 6 months, 1 year, and yearly to 5 years
Binary restenosis in both in-stent and in-segment | at 9 month angiographic follow-up
Graft patency and reocclusion rate | at 9 months angiographic follow-up
Late luminal loss in both in-stent and in-segment | at 9 month angiographic follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Seung-Jung Park, MD, PhD, Principal Investigator — Department of Medicine, Asan Medical Center, University of Ulsan College of Medicine
Locations (13):
- South Korea (13):
  - Daegu Catholic University Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - St.Mary's Catholic Medical Center, Seoul
  - Yonsei University Medical Center, Seoul
  - Ajou University Hospital, Suwon
  - Ulsan University Hospital, Ulsan

REFERENCES:
- [Derived] Gaba P, Sabik JF, Murphy SA, Bellavia A, O'Gara PT, Smith PK, Serruys PW, Kappetein AP, Park SJ, Park DW, Christiansen EH, Holm NR, Nielsen PH, Sabatine MS, Stone GW, Bergmark BA. Percutaneous Coronary Intervention Versus Coronary Artery Bypass Grafting in Patients With Left Main Disease With and Without Diabetes: Findings From a Pooled Analysis of 4 Randomized Clinical Trials. Circulation. 2024 Apr 23;149(17):1328-1338. doi: 10.1161/CIRCULATIONAHA.123.065571. Epub 2024 Mar 11. PMID 38465592
- [Derived] Kim TO, Kang DY, Ahn JM, Kim MJ, Lee PH, Kim H, Choi Y, Lee J, Lee JM, Jo HH, Park YS, Lim SM, Park SJ, Park DW. Impact of Target Lesion Revascularization on Long-Term Mortality After Percutaneous Coronary Intervention for Left Main Disease. JACC Cardiovasc Interv. 2024 Jan 8;17(1):32-42. doi: 10.1016/j.jcin.2023.10.068. PMID 38199751
- [Derived] Gaba P, Christiansen EH, Nielsen PH, Murphy SA, O'Gara PT, Smith PK, Serruys PW, Kappetein AP, Park SJ, Park DW, Stone GW, Sabik JF, Sabatine MS, Holm NR, Bergmark BA. Percutaneous Coronary Intervention vs Coronary Artery Bypass Graft Surgery for Left Main Disease in Patients With and Without Acute Coronary Syndromes: A Pooled Analysis of 4 Randomized Clinical Trials. JAMA Cardiol. 2023 Jul 1;8(7):631-639. doi: 10.1001/jamacardio.2023.1177. PMID 37256598
- [Derived] Kim T, Kang DY, Kim S, Lee JH, Kim AR, Lee Y, Oh HJ, Jang M, Lee J, Kim JH, Lee PH, Ahn JM, Park SJ, Park DW; PRECOMBAT Extended Study Investigators. Impact of Complete or Incomplete Revascularization for Left Main Coronary Disease: The Extended PRECOMBAT Study. JACC Asia. 2023 Jan 24;3(1):65-74. doi: 10.1016/j.jacasi.2022.10.007. eCollection 2023 Feb. PMID 36873760
- [Derived] Jeong YJ, Ahn JM, Hyun J, Lee J, Kim JH, Yang Y, Choe K, Park H, Kang DY, Lee PH, Kang SJ, Lee SW, Kim YH, Lee CW, Park SW, Park SJ, Park DW. Ten-year Outcomes After Drug-Eluting Stents or Bypass Surgery for Left Main Coronary Disease in Patients With and Without Diabetes Mellitus: The PRECOMBAT Extended Follow-Up Study. J Am Heart Assoc. 2021 Jul 20;10(14):e019834. doi: 10.1161/JAHA.120.019834. Epub 2021 Jul 9. PMID 34238026
- [Derived] Park DW, Ahn JM, Park H, Yun SC, Kang DY, Lee PH, Kim YH, Lim DS, Rha SW, Park GM, Gwon HC, Kim HS, Chae IH, Jang Y, Jeong MH, Tahk SJ, Seung KB, Park SJ; PRECOMBAT Investigators. Ten-Year Outcomes After Drug-Eluting Stents Versus Coronary Artery Bypass Grafting for Left Main Coronary Disease: Extended Follow-Up of the PRECOMBAT Trial. Circulation. 2020 May 5;141(18):1437-1446. doi: 10.1161/CIRCULATIONAHA.120.046039. Epub 2020 Mar 30. PMID 32223567
- [Derived] Sotomi Y, Onuma Y, Cavalcante R, Ahn JM, Lee CW, van Klaveren D, de Winter RJ, Wykrzykowska JJ, Farooq V, Morice MC, Steyerberg EW, Park SJ, Serruys PW. Geographical Difference of the Interaction of Sex With Treatment Strategy in Patients With Multivessel Disease and Left Main Disease: A Meta-Analysis From SYNTAX (Synergy Between PCI With Taxus and Cardiac Surgery), PRECOMBAT (Bypass Surgery Versus Angioplasty Using Sirolimus-Eluting Stent in Patients With Left Main Coronary Artery Disease), and BEST (Bypass Surgery and Everolimus-Eluting Stent Implantation in the Treatment of Patients With Multivessel Coronary Artery Disease) Randomized Controlled Trials. Circ Cardiovasc Interv. 2017 May;10(5):e005027. doi: 10.1161/CIRCINTERVENTIONS.117.005027. PMID 28495897
- [Derived] Sotomi Y, Cavalcante R, van Klaveren D, Ahn JM, Lee CW, de Winter RJ, Wykrzykowska JJ, Onuma Y, Steyerberg EW, Park SJ, Serruys PW. Individual Long-Term Mortality Prediction Following Either Coronary Stenting or Bypass Surgery in Patients With Multivessel and/or Unprotected Left Main Disease: An External Validation of the SYNTAX Score II Model in the 1,480 Patients of the BEST and PRECOMBAT Randomized Controlled Trials. JACC Cardiovasc Interv. 2016 Aug 8;9(15):1564-72. doi: 10.1016/j.jcin.2016.04.023. PMID 27491605
- [Derived] Ahn JM, Roh JH, Kim YH, Park DW, Yun SC, Lee PH, Chang M, Park HW, Lee SW, Lee CW, Park SW, Choo SJ, Chung C, Lee J, Lim DS, Rha SW, Lee SG, Gwon HC, Kim HS, Chae IH, Jang Y, Jeong MH, Tahk SJ, Seung KB, Park SJ. Randomized Trial of Stents Versus Bypass Surgery for Left Main Coronary Artery Disease: 5-Year Outcomes of the PRECOMBAT Study. J Am Coll Cardiol. 2015 May 26;65(20):2198-206. doi: 10.1016/j.jacc.2015.03.033. Epub 2015 Mar 15. PMID 25787197
- [Derived] Park SJ, Kim YH, Park DW, Yun SC, Ahn JM, Song HG, Lee JY, Kim WJ, Kang SJ, Lee SW, Lee CW, Park SW, Chung CH, Lee JW, Lim DS, Rha SW, Lee SG, Gwon HC, Kim HS, Chae IH, Jang Y, Jeong MH, Tahk SJ, Seung KB. Randomized trial of stents versus bypass surgery for left main coronary artery disease. N Engl J Med. 2011 May 5;364(18):1718-27. doi: 10.1056/NEJMoa1100452. Epub 2011 Apr 4. PMID 21463149